CLINICAL TRIAL: NCT00250978
Title: Phase I of Bevacizumab Plus Chemotherapy in Patients With Malignant Pleural Effusion Due to Advanced Non-Small Cell Lung Cancer
Brief Title: Ph I:Bevacizumab + Chemotherapy in Pts w/Malig Pleural Effusion Due to Adv NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Christopher Azzoli, MD, Memorial Sloan Kettering Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-089
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Advanced Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Drug Therapy

INTERVENTIONS:
Drug: bevacizumab with chemotherapy, Pleur-XTM catheter placement — After Pleur-XTM catheter placement patients will receive bevacizumab 15mg/kg IV x 1 dose as a single agent.Three weeks later, chemotherapy will be initiated according to routine clinical practice along with continued use of bevacizumab.

SUMMARY:
Your lung cancer has caused fluid to build up in the space around your lung. This fluid is called a malignant pleural effusion. This fluid takes up space in your chest, and prevents your lung from fully filling with air. As a result, you may be experiencing shortness of breath, cough, or chest discomfort. Your doctors have determined that you would feel better if a surgeon or pulmonary specialist removed this fluid immediately. Your doctors are offering to admit you to the hospital, and drain the fluid using a Pleur-XTM catheter.

Once the Pleur-X catheter is in place, your doctors would like to start your chemotherapy.

Your doctors have decided to treat you with chemotherapy. If the chemotherapy works to kill the cancer cells in your body, the cancer will make less fluid, and your doctors will be able to remove the Pleur-XTM catheter sooner.

It is possible that adding a second drug to the chemotherapy, called bevacizumab may make he fluid dry up even faster. It is not known whether adding bevacizumab to chemotherapy for patients with a Pleur-XTM catheter in place is more helpful, or potentially more harmful, than using chemotherapy alone. For this reason, only patients enrolled in this research protocol can receive both chemotherapy and bevacizumab while they have a Pleur-XTM catheter in place.

The purpose of this research study is to determine whether chemotherapy may be delivered safely with a Pleur-XTM catheter in place.

DETAILED DESCRIPTION:
The study will be conducted in patients with advanced NSCLC (stage IIIB-IV) who have MPE requiring therapeutic drainage, and are also eligible for treatment with chemotherapy plus bevacizumab (as defined in protocol Section 6.0). All patients will undergo placement of a Pleur-XTM catheter as part of routine practice. Eligible patients may enroll in the protocol prior to, or within 10 days following placement of their Pleur-XTM catheter. Upon enrollment, patients will be given a logsheet on which to record the volume of pleural fluid drained from their catheter. Only patients who, in the opinion of the treating physician, do not have a hemorrhagic pleural effusion (grossly bloody, or pleural fluid hemoglobin concentration > 25% of blood hemoglobin concentration) may remain on study. In addition, only patients who, in the opinion of the treating physician, have satisfactory placement of their Pleur-XTM catheter may remain on study.

Approximately 15 patients will be enrolled with the goal to treat 10 patients with chemotherapy plus bevacizumab. The additional enrollments will be necessary in that it is estimated that approximately 1 in 3 patients will be taken off study due to failure of Pleur-XTM catheter placement, or discovery of hemorrhagic effusion.

Patients who remain on study will begin chemotherapy. All eligible patients will receive bevacizumab 15mg/kg IV x 1 dose as a single agent. Three weeks later, chemotherapy will be initiated according to routine clinical practice along with continued use of bevacizumab. Acceptable chemotherapy regimens for this protocol are detailed in Section 5.0 of the protocol. Only the administration of bevacizumab will be governed by the protocol (Section 11.0). Dose reductions of all other drugs will be made according to routine clinical practice. Pleural fluid will be drained from the Pleur-XTM at least every other day (qod), and volume recorded by the patient in a log book. Pleur-XTM catheters may be removed when pleural symphysis is achieved (defined in Section 12.0), or at the discretion of the treating physician. The schedule of follow-up visits may vary according to the chemotherapy regimen, however all patients must be evaluated in the clinic at least every 3 weeks with a doctor visit to record drainage volume, and status of their Pleur-XTM catheter.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with pathologically confirmed stage IIIB-IV non-small cell lung cancer who are eligible for systemic chemotherapy, and also have a malignant pleural effusion which requires therapeutic drainage.
* Karnofsky performance status >=70%
* Adequate coagulation studies, blood counts, renal and hepatic function:

aPTT < 33.8 seconds, PT/INR < 1.12, WBC >= 3,000/ul, hemoglobin >= 9.0 g/dl, platelet count >=100,000/ul, total bilirubin <= 1.3 mg/dl, AST/ALT <= 2.0 X UNL, Alk Phos <= 2.5 X UNL, creatinine <= 1.5 mg/dl

* Ability to maintain a Pleur-XTM drainage catheter
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Exclusion Criteria:

* Prior bevacizumab
* Squamous cell histology
* Hemoptysis within the past 3 months that brings up more than 1/2 teaspoon of red blood
* Patients already known to have hemorrhagic pleural effusion, defined as a grossly bloody pleural effusion in the opinion of the treating physician,or pleural fluid hemoglobin concentration >= 25% of blood hemoglobin concentration .
* Known brain metastases
* Clinically significant cardiovascular disease, uncontrolled hypertension, or peripheralvascular disease
* History of cerebrovascular accident or transient ischemic attack within the past six months
* Pregnancy
* Urine protein: creatinine (UPC) ratio >= 1.0 at screening
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0
* History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 28 days prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Patients must not be receiving daily treatment with aspirin (>= 325 mg/day) or daily use of non-steroidal anti-inflammatory agents known to inhibit platelet function including ibuprofen, dipyridamole, ticlopidine, clopidogrel and/or cilostazol.
* Patients must not be on therapeutic anticoagulation with warfarin, heparin or low molecular weight heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety and feasibility of administering chemotherapy plus bevacizumab to patients with metastatic NSCLC and MPE following insertion of a Pleur-XTM catheter. | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G. Azzoli, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org